CLINICAL TRIAL: NCT00078689
Title: Combination Daclizumab/Sirolimus Therapy For the Induction of Immune Tolerance in Non-Infectious Intermediate and Posterior Uveitis
Brief Title: Daclizumab and Sirolimus to Treat Uveitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040115; 04-EI-0115
Record Dates: First submitted 2004-03-04; First posted 2004-03-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-18

CONDITIONS: Uveitis
Keywords: Sirolimus; Daclizumab; Inflammation; Induce Tolerance; Uveitis; Immune Tolerance; T Cell
MeSH Terms: conditions — Uveitis; Inflammation | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This study will examine whether the combination of the drugs daclizumab and sirolimus can effectively treat adults with uveitis, an eye inflammation. Daclizumab is a monoclonal antibody that is designed to prevent a specific chemical interaction needed for immune cells called lymphocytes to produce inflammation. Sirolimus is an immune-suppressing drug that also controls lymphocyte activity and is marketed to prevent organ rejection in kidney transplants.

Patients 18 years of age and older with non-infectious uveitis in one or both eyes who are being treated with daclizumab and have not had a relapse or disease flare for 6 months before entering this trial may be eligible for this study. Candidates are screened with a medical history and physical examination, blood tests, complete eye examination, and pregnancy test for women who can have children. Women of child-bearing potential who enroll in this study will have a pregnancy test every 12 weeks.

After enrollment, participants have the following additional exams:

* Fluorescein angiography: This test is done to check for abnormalities of eye blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken with a special camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible abnormalities. This test is done at enrollment and after 1 year, unless additional tests are needed for medical management.
* Pelvic ultrasound and urine test: These tests are done at enrollment and after 1 year to check the kidneys, lymph nodes, and pelvic area.
* Blood tests: Blood tests are done at enrollment and every 3 to 6 months for laboratory and immunology study

Patients receive daclizumab subcutaneously (under the skin) or in infusions at regularly scheduled visits for 52 weeks. At each treatment, blood pressure, pulse, breathing rate, and temperature are monitored. After the first 52 weeks, patients whose disease remains quiet increase the time between injections to 6 weeks and then to 8 weeks. Patients who are doing well at this time may stop daclizumab.

One or 2 days after the first daclizumab treatment, patients receive 6 mg of sirolimus by mouth. Their blood pressure, pulse, breathing rate, and temperature are monitored for at least 60 minutes. Two days after the first dose, patients begin 2-mg maintenance doses every other day for 2 weeks. If there are no intolerable side effects, the dose is increased to 2 mg daily for the next 2 weeks. Patients who have no intolerable side effects at that dose continue the medication for another 4 weeks. Patients who experience intolerable side effects may decrease the medication to every other day or withdraw from the study. After week 78 of the study, if the daclizumab treatments are stopped, the sirolimus dose is reduced within 8 weeks and may eventually be discontinued if the patient continues to do well.

Patients who experience any of the following will leave the study:

* Inflammation flare that requires concomitant treatment with additional systemic immunosuppressive medications, such as prednisone or cyclosporine
* Disease flares more than twice in the first year
* Any disease flares in the second year

DETAILED DESCRIPTION:
We propose to investigate the possible efficacy of combination daclizumab and sirolimus therapy to induce peripheral immune tolerance in participants presenting with non-infectious intermediate and posterior uveitis. This will be performed using a Phase I/II pilot study. Subjects on daclizumab monotherapy will receive a 6 mg loading dose of oral sirolimus at week 0, followed by a 2 mg dose every other day for 2 weeks. If tolerated, the subject will be increased to a 2 mg daily dose. After one year of combination therapy, the subject will be tapered off daclizumab first and then sirolimus. The primary outcome will be the ability of the participant to be successfully tapered off daclizumab and sirolimus while their disease remains quiet (vitreous haze less than or equal to Trace) for 24 weeks on no systemic immunosuppressive medications (approximately week 134).

ELIGIBILITY:
* INCLUSION CRITERIA:

Participant is 18 years of age or older.

Participant with uveitis in one or both eyes on daclizumab monotherapy without disease flare in the past 6 months.

Participant agrees to use acceptable birth control methods throughout the course of the study and for 6 months after completion of treatment with daclizumab or sirolimus.

Participant is able to understand and sign a consent form before entering the study.

EXCLUSION CRITERIA:

Participant with a history of hypersensitivity to FK506 or sirolimus.

Participant who has had major surgery in the past 6 months.

Participant is pregnant or lactating.

Participant with active chronic or acute infections.

Participant with malignancy other than squamous cell carcinoma in situ.

Participant with uncontrolled hyperlipidemia at the time of enrollment.

Participant without VZV antibodies.

Participant without Hepatitis antibodies (anti-HAV or anti-HBc) AND with any one of the following risk factors for acquiring hepatitis: IV drug abuse, male homosexual activity, hemophilia, prostitution, or health care work.

Participant requiring systemic anti-fungal therapy with ketoconazole for whom no other acceptable alternative anti-fungal therapy exists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2004-03-03; Study Completion 2008-07-18

PRIMARY OUTCOMES:
Ability to taper off drug while disease remains quiet at week 108 while receiving no concomitant systemic immunosuppressive medications.

SECONDARY OUTCOMES:
Number and severity of disease flares requiring changes in concomitant immunosuppressive medication.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Caspi RR, Roberge FG, McAllister CG, el-Saied M, Kuwabara T, Gery I, Hanna E, Nussenblatt RB. T cell lines mediating experimental autoimmune uveoretinitis (EAU) in the rat. J Immunol. 1986 Feb 1;136(3):928-33. PMID 2416842
- [Background] Ramos EL, Leggat JE, Milford EL, Kirkman RL, Tilney NL, Strom TB, Shapiro ME, Waldmann TA, Carpenter CB. In vivo anti-interleukin-2 receptor (anti-Tac) therapy is immunosuppressive, but not tolerogenic. Trans Assoc Am Physicians. 1989;102:231-9. No abstract available. PMID 2534707
- [Background] Herve P, Wijdenes J, Bergerat JP, Bordigoni P, Milpied N, Cahn JY, Clement C, Beliard R, Morel-Fourrier B, Racadot E, et al. Treatment of corticosteroid resistant acute graft-versus-host disease by in vivo administration of anti-interleukin-2 receptor monoclonal antibody (B-B10). Blood. 1990 Feb 15;75(4):1017-23. PMID 2136244